CLINICAL TRIAL: NCT06504056
Title: Risk Stratification and Early Prevention Strategies for Non-compaction of Ventricular Myocardium (CAPTAIN): a Multicenter, Retrospective-prospective, Cohort Study
Brief Title: Risk Stratification and Early Prevention Strategies for Non-compaction of Ventricular Myocardium (CAPTAIN)
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2024LSYY-053
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Isolated Noncompaction of the Ventricular Myocardium
Keywords: Isolated Noncompaction of the Ventricular Myocardium; Prognostic factors
MeSH Terms: conditions — Isolated Noncompaction of the Ventricular Myocardium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — For the retrospectively enrolled patients, the investigators will collect their biological samples previously housed in the Biobank of The First Affiliated Hospital of Xi'an Jiaotong University.
  For the prospectively enrolled patients, the investigators will collect a variety of biological samples at admission, before discharge, 1st, 3rd, 6th, 9th month, 1st, 2nd, 3rd year after discharge, including blood, urine, feces, other types of body fluids (such as pericardial effusion), tissue samples from surgery and biopsy (such as pericardial effusion, myocardial tissue, tumors, blood clots, etc.), or samples that need to be disposed of as medical waste (blood clots, etc.), or the sample itself requires pathological examination to assist in diagnosis and treatment (e.g. endocardial muscle biopsy).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Left ventricle group: The patients mainly had thickened myocardial wall with a thin, compacted epicardial layer and a thicker endocardial layer, and were diagnosed with LVNC.
  Interventions: Biological: Diagnosis of NVM
- Right ventricle group: The patients mainly had thickened myocardial wall with a thin, compacted epicardial layer and a thicker endocardial layer, and were diagnosed with right NVM.
  Interventions: Biological: Diagnosis of NVM
- Two sided ventricle group: The patients mainly had thickened myocardial wall with a thin, compacted epicardial layer and a thicker endocardial layer, and were diagnosed with right and left ventricle NVM.
  Interventions: Biological: Diagnosis of NVM

INTERVENTIONS:
Biological: Diagnosis of NVM — The term 'left ventricular non-compaction' (LVNC) has been used to describe a ventricular phenotype characterized by prominent LV trabeculae and deep intertrabecular recesses. The myocardial wall is often thickened with a thin,compacted epicardial layer and a thickened myocardial layer. In some patients, this abnormal trabecular architecture is associated with LV dilatation and systolic dysfunction. Left ventricular non-compaction is frequently a familial trait and is associated with variants in a range of genes, including those encoding proteins of the sarcomere, Z-disc, cytoskeleton, and nuclear envelope.
  Groups: Left ventricle group
Biological: Diagnosis of NVM — The term 'left ventricular non-compaction' (LVNC) has been used to describe a ventricular phenotype characterized by prominent LV trabeculae and deep intertrabecular recesses. The myocardial wall is often thickened with a thin,compacted epicardial layer and a thickened myocardial layer. In some patients, this abnormal trabecular architecture is associated with LV dilatation and systolic dysfunction. Left ventricular non-compaction is frequently a familial trait and is associated with variants in a range of genes, including those encoding proteins of the sarcomere, Z-disc, cytoskeleton, and nuclear envelope.
  Groups: Right ventricle group
Biological: Diagnosis of NVM — The term 'left ventricular non-compaction' (LVNC) has been used to describe a ventricular phenotype characterized by prominent LV trabeculae and deep intertrabecular recesses. The myocardial wall is often thickened with a thin,compacted epicardial layer and a thickened myocardial layer. In some patients, this abnormal trabecular architecture is associated with LV dilatation and systolic dysfunction. Left ventricular non-compaction is frequently a familial trait and is associated with variants in a range of genes, including those encoding proteins of the sarcomere, Z-disc, cytoskeleton, and nuclear envelope.
  Groups: Two sided ventricle group

SUMMARY:
This study intends to retrospectively-prospectively enroll NVM patients from multiple centers to establish a natural population cohort of NVM patients. By collecting clinical data and biological samples from surgical patients, the investigators will construct a prognosis prediction system for NVM, optimize risk stratification, explore new strategies for the early prevention and treatment of NVM, and improve the efficiency of clinical treatment of NVM patients.

DETAILED DESCRIPTION:
This study intends to retrospectively-prospectively enroll NVM patients from multiple centers to establish a natural population cohort of NVM patients. By collecting clinical data and biological samples from surgical patients, the investigators will construct a prognosis prediction system for NVM, optimize risk stratification, explore new strategies for the early prevention and treatment of NVM, and improve the efficiency of clinical treatment of NVM patients.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of nvm was confirmed by cardiac ultrasound, electrocardiogram, magnetic resonance angiography, pathological examination and gene sequencing.
* Patients or their families agreed to participate in the study and authorized informed consent.

Exclusion Criteria:

* Incomplete clinical data.
* Do not agree to the inclusion or refuse to authorize the informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with NVM at all centers including The First Affiliated Hospital of Xi'an Jiaotong University.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in the incidence of mortality rate | At diagnosis, before discharge (about 7 days), 1, 3, 6, 9 month, 1, 2, 3 year.
  The survival status will be obtained from the medical records and phone calls to patients or their family members.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yan, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiantong University, Xi'an, Shaanxi, China